CLINICAL TRIAL: NCT03763539
Title: Ultraslow Full-power SWL Versus Slow Power-ramping SWL in Stones With High Attenuation Value
Acronym: SWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSheemy, Associate Professor of Urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5124
Record Dates: First submitted 2018-12-01; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Renal Stones
Keywords: renal stones; SWL; High density stones; Ultraslow SWL; Slow SWL; Ramping; Pause
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultraslow shock wave lithotripsy (SWL) (Active Comparator): SWL at ultraslow rate of 30 SW/min. Power ramping at the first 100 SW from 6 to 18 kv followed by safety pause for two minutes then power ramping from 18 to 22kv during the second 100 SW followed by safety pause for another two minutes.
  The rest of the session at 22kv (full power).
  Interventions: Procedure: SWL
- Slow power-ramping SWL (Active Comparator): SWL at a slow rate of 60 SW/min. Power ramping from 6 - 10 kv during the first 500 SW then from 11 - 14 kv during the second 500 SW then from 15 - 18 kv during the following 500 SW then from 19 - 22 kv during the remaining 1000 - 1500 SW.
  Interventions: Procedure: SWL

INTERVENTIONS:
Procedure: SWL — Shock wave lithotripsy
  Other Names: ESWL

SUMMARY:
Ultraslow full-power SWL versus slow power-ramping SWL in stones with high attenuation value

DETAILED DESCRIPTION:
To evaluate the efficacy of ultraslow rate of SWL versus slow rate, power ramping SWL.

ELIGIBILITY:
Inclusion Criteria:

* single renal stone less than or equal to 3 cm (2 cm for lower calyceal stones)
* radio-opaque stone
* high attenuation value (≥ 1000 HU) stone

Exclusion Criteria:

* Abnormal renal anatomy
* renal insufficiency
* solitary kidney
* coagulopathies
* uncontrolled hypertension
* renal artery or aortic aneurysm
* active urinary tract infection
* pregnancy
* severe skeletal malformations (spinal deformity) precluding proper stone localization
* skin to stone distance (SSD) > 11 cm
* BMI > 30 Kgm/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
stone free rate | 3 months following last session of SWL
  Complete clearance of stones in addition to clinically insignificant residual fragments

SECONDARY OUTCOMES:
Complications | 1 year following last session of SWL
  Comparison of complications in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Aref Al-Dessoukey, Ass. Prof., Study Director — Beni-Suef University
Locations (1):
- Beni-Suef Hospitals, Banī Suwayf, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03763539/SAP_000.pdf